CLINICAL TRIAL: NCT00972231
Title: Iron Overload and Growth Velocity in Thalassemia and Sickle Cell Anemia
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Hematology Unit and Pediatric Dpt B, HaEmek Medical Center, Israel
Other Study IDs: 0133-08-EMC
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Thalassemia; Sickle Cell Disease
Keywords: Thalassemia Major; Thalassemia Intermedia; Sickle Cell Anemia; Sickle Cell Thalassemia; Iron Overload; Growth Velocity
MeSH Terms: conditions — Thalassemia; Anemia, Sickle Cell; beta-Thalassemia; Iron Overload

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Thalassemia Group: Patients suffering from Thalassemia Major and patients with Thalassemia Intermedia
  Interventions: Other: Medical Chart Summary
- Sickle Cell Group: Patients with Sickle Cell Anemia and Sickle Cell Thalassemia
  Interventions: Other: Medical Chart Summary

INTERVENTIONS:
Other: Medical Chart Summary — Summary of the Medical Files including annual growth velocity, endocrine function and iron overload status.

SUMMARY:
Iron overload impaired growth in Thalassemia patients due to iron deposition in the endocrine glands, including the hypophysis and gonads. The issue of iron overload in Sickle Cell Anemia is recently studied more extensively and preliminary studies shows that endocrine damage is rarer in those patients.

Growth velocity was not systematically studied in patients with Iron Overload, even in thalassemia patients in spite several studies that assess the endocrine function in those patients. In Sickle Cell Patients this issue was not studied.

The purpose of this study is to assess the growth velocity in a cohort of Thalassemia Major and Intermedia patients and compare the results to another group of Sickle Cell patients, including Sickle cell thalassemia.

DETAILED DESCRIPTION:
Growth velocity, endocrine function and iron overload status will be studied in the patients that are in follow up at the Pediatric Hematology Unit, at the Ha'Emek Medical Center.

Patients who were lost from follow up or insufficient data about growth in the past will not included in the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients in follow up with available medical charts.

Exclusion Criteria:

* Patients lost from follow up or without enough data to calculate growth velocity or clinical and laboratory endocrine assessment or missing data about iron status.

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 150 patients suffering from hemoglobinopathies are treated at the Pediatric Hematology Unit, Ha'Emek Medical Center. This include Thalassemia Major blood transfused and treated by chelators, Thalassemia Intermedia patients ussualy not transfused, some of them treated by Hydroxyurea, and two groups of Sickle cell patients, Sickkle cell homozygous and Sickle cell thalassemia. Most of the Sickle cell patients are treated with Hydroxyurea.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Iron Overload and Growth Velocity in Thalassemia and Sickle Cell Anemia | One year
  Analysis of Growth Velocity in Thalassemia and Sickle Cell Anemia and correlation with Iron Overload

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Principal Investigator — Pediatric Dpt B and Pediatric Hemaology Unit - Ha'Emek Medical Center - Afula - Israel; Carina Levin, MD, Principal Investigator — Pediatric Hematology Unit, Ha'Emek Medical Center, Afula, Israel; Daniela Mathov, Student, Principal Investigator — Pediatic Hematology Unit, Ha'Emek Medical Center, Afula, Israel
Locations (1):
- Pediatric Hematology Unit - Ha'Emek Medical Center, Afula, Afula, Israel